CLINICAL TRIAL: NCT05665855
Title: The Effects of Acute Ketone Monoester Supplementation on Exercise Efficiency and the Influence of Dose and Intensity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Martin Gibala, Principal Investigator, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15110
Record Dates: First submitted 2022-11-17; First posted 2022-12-27 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Exercise; Ketosis
Keywords: Efficiency
MeSH Terms: conditions — Motor Activity; Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone higher dose (Experimental): An acute bout of exercise performed after the ingestion of a commercial supplement intended to provide ~0.6 g of ketone monoester per kg body mass of the participant.
  Interventions: Dietary Supplement: Ketone monoester
- Ketone lower dose (Experimental): An acute bout of exercise performed after the ingestion of a commercial supplement intended to provide ~0.3 g of ketone monoester per kg body mass of the participant.
  Interventions: Dietary Supplement: Ketone monoester
- Control (Placebo Comparator): An acute bout of exercise performed after the ingestion of a taste-matched placebo supplement.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone monoester — A commercial liquid ketone monoester supplement.
  Arms: Ketone higher dose; Ketone lower dose
Other: Placebo — A liquid placebo that is taste-matched to the ketone monoester supplement.
  Arms: Control

SUMMARY:
Diet can alter blood ketone levels and this in turn may affect exercise capacity. This study will determine if the acute ingestion of a ketone supplement alters cycling exercise efficiency. Participants will perform three trials in a randomized order. Each trial will involve an incremental exercise protocol on a stationary cycle ergometer to volitional fatigue. Participants will ingest either a high or low dose of a ketone supplement or a taste-matched placebo drink prior to exercise. Blood samples will be obtained to assess selected metabolic responses. This study will provide information regarding the effect of ketone supplementation on exercise efficiency.

DETAILED DESCRIPTION:
This study will determine if the acute ingestion of a ketone supplement alters cycling exercise efficiency. Trained participants with cycling experience will be recruited. Participants will perform three trials in a randomized order. Each trial will involve a 3-minute warm-up followed by an incremental ramp test. The ramp will initially consist of three, 5-minute stages performed at relative workloads corresponding to 75%, 100%, and 125% of individual ventilatory threshold intensity. This will be followed by a further incremental ramp test to volitional fatigue. Participants will ingest either a high or low dose of a ketone supplement or a taste-matched placebo drink prior to exercise using a randomized, double-blind crossover design. Diet prior to exercise will be standardized between trials for a given participant. Blood samples will be obtained to assess selected metabolic responses. This study will provide information regarding the effect of ketone supplementation on exercise efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Be habitually consuming ≥50 g/d of carbohydrate (i.e., not following a ketogenic diet).
* Be engaged in endurance-type exercise >3h/wk.
* Have an estimated VO2peak of ≥90% for age and sex as estimated by an online calculator found at www.worldfitnesslevel.org.

Exclusion Criteria:

* Experiencing a condition that might preclude safe participation in physical activity and exercise, as determined by answering "Yes" to any question on Page 1 of the Canadian Society for Exercise Physiology Get Active Questionnaire.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Exercise efficiency | Continuous measurement made over each of three, 5-minute consecutive stages of an incremental cycle exercise test at relative workloads corresponding to 75%, 100%, and 125% of individual ventilatory threshold intensity
  Power output expressed relative to pulmonary oxygen uptake to determine cycling economy in watt per litre of oxygen per minute

SECONDARY OUTCOMES:
Heart rate | Continuous measurement made over each of three, 5-minute consecutive stages of an incremental cycle exercise test at relative workloads corresponding to 75%, 100%, and 125% of individual ventilatory threshold intensity
  Mean heart rate
Rating of perceived exertion | Measurement made at the end of each of three, 5-minute consecutive stages of an incremental cycle exercise test at relative workloads corresponding to 75%, 100%, and 125% of individual ventilatory threshold intensity
  Rating of perceived exertion measured using a 6-20 scale
Ketone body content in venous blood | Measurement made immediately prior to exercise
  Mixed venous blood content of the ketone body beta-hydroxybutyrate

CONTACTS AND LOCATIONS:
Overall Officials: Martin J Gibala, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No